CLINICAL TRIAL: NCT06975592
Title: Study on the Mechanism of Multi-group Analysis of the Influence of Depression on Common Cardiovascular Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Depression and CVD
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Depression and CVD
Keywords: Depression and cardiovascular diseases
MeSH Terms: conditions — Depression; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples of feces, urine, peripheral blood and oral secretions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy control group: 1) Good health and no gastrointestinal diseases; 2) No previous history of mental illness; 2) No previous history of cardiovascular disease;
- Depression group: 1. Meet the diagnostic criteria of the latest guidelines for depression, and be clinically diagnosed by at least two psychiatrists;
  2. Patients with first-episode depression;
  3. Have not taken any psychoactive drugs before or have not taken any psychoactive drugs within 4 weeks.
- Depression with cardiovascular disease group: 1. Meet the diagnostic criteria of the latest guidelines for depression, and be clinically diagnosed by at least two psychiatrists;
  2. Patients with first-episode depression;
  3. Have not taken any psychoactive drugs before or have not taken any psychoactive drugs within 4 weeks.
  4. There is definite clinical evidence of heart failure, coronary heart disease, hypertension or arrhythmia.

SUMMARY:
Cardiovascular disease is the main cause of death in the world, accounting for 32% of all deaths. In 2019, the number of people suffering from cardiovascular diseases in the world was about 523 million, of which about 18.6 million died of cardiovascular diseases. Although great progress has been made in reducing the burden of cardiovascular diseases by controlling typical risk factors, there is still a lack of effective intervention means and measures for cardiovascular diseases induced by atypical risk factors (such as environmental pollution, obesity and anxiety and depression).

Depression is a health problem as common as cardiovascular disease, and it has been proved to be an important risk factor of cardiovascular disease. Previous studies have shown that depression is related to the increased risk of subsequent cardiovascular events, including myocardial infarction, angina pectoris, stroke and cardiovascular mortality. The risk of cardiovascular disease in patients with major depression is about 72% higher than that in healthy control group.

Previous studies have shown that compared with healthy people, the intestinal microbial composition of patients with major depression, especially the microbial diversity and the relative abundance of specific bacterial groups, has changed significantly. Many studies have also confirmed that dysbacteriosis may be an important cause of MDD, and with the passage of time, the pathological changes caused by MDD will further destroy the intestinal environment and lead to dysbacteriosis. In addition, intestinal microflora can also produce a variety of important mediators, such as metabolites produced by bacterial fermentation of food, host molecules modified by bacteria (bile acids, etc.) or direct products of bacteria, which also play an important role in the pathogenesis of MDD. In recent years, both population studies and animal experiments have found that the changes in the composition and function of intestinal flora (that is, the imbalance of intestinal microbial flora) will accelerate the occurrence and development of cardiovascular diseases. Intestinal flora will metabolize the food ingested by the host into a series of metabolites, including trimethylamine oxide, short-chain fatty acids, secondary bile acids and indole sulfate, etc. These metabolites will affect the physiological process of the host by activating various signal pathways, thus affecting the occurrence and development of cardiovascular diseases (such as coronary heart disease, hypertension, arrhythmia and heart failure).

All the above results suggest that intestinal flora and its metabolites play an important role in promoting the occurrence and development of cardiovascular diseases in depression, but its internal mechanism is not completely clear. Therefore, it is of great significance to deeply explore the pathophysiological mechanism of depression on cardiovascular diseases for guiding the prevention and treatment of cardiovascular diseases.

A total of 300 people were enrolled in this study, which were divided into healthy control group, depression group and depression combined with cardiovascular disease group, with 100 cases in each group. Samples of patients' feces, urine peripheral blood and oral secretions were collected and analyzed by multi-omics. Subsequently, after 6 months, 1 year, 2 years and 5 years after discharge, the clinical prognosis of the patients was obtained and recorded.

The purpose of this study is to discover and deeply explore the pathophysiological mechanism of depression on common cardiovascular diseases (coronary heart disease, hypertension, arrhythmia or heart failure) through the research methods of 16S rDNA sequencing, metagenome sequencing and metabonomics, so as to provide theoretical basis for comprehensive treatment of cardiovascular diseases caused by depression, and at the same time provide potential biomarkers and prevention targets for cardiovascular diseases caused by depression.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy control group 1) Good health and no gastrointestinal diseases; 2) No previous history of mental illness; 3) No previous history of cardiovascular disease;
2. Depression group

1) Meet the diagnostic criteria of the latest guidelines for depression, and be clinically diagnosed by at least two psychiatrists; 2) Patients with first-episode depression; 3) Have not taken any psychoactive drugs before or have not taken any psychoactive drugs within 4 weeks.

3. Depression with cardiovascular disease group

1. Meet the diagnostic criteria of the latest guidelines for depression, and be clinically diagnosed by at least two psychiatrists;
2. Patients with first-episode depression;
3. Have not taken any psychoactive drugs before or have not taken any psychoactive drugs within 4 weeks.
4. There is definite clinical evidence of heart failure, coronary heart disease, hypertension or arrhythmia.

Exclusion Criteria:

1. Have a history of alcohol dependence, organic brain diseases, nervous system diseases and other complex mental diseases;
2. Long-term use of psychoactive drugs/use of psychoactive drugs within 4 weeks;
3. Patients with thyroid dysfunction
4. Patients with severe liver and kidney dysfunction;
5. Patients with chronic obstructive pulmonary disease, interstitial pulmonary fibrosis and pulmonary hypertension;
6. Patients with autoimmune diseases and tumors;
7. used antibiotics, yogurt or other drugs or foods that affect intestinal flora within 4 weeks;
8. Pregnant or lactating women;
9. There is a serious impairment of cognitive function, which makes it impossible to cooperate with the research procedure;
10. Have received invasive medical procedures such as gastroscopy and colonoscopy in the past three months;
11. The diet has changed greatly in the past week;
12. Participate in simultaneous clinical trials;
13. Refuse to sign the informed consent for participating in the experiment.

Max Age: 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Samples of feces, urine and peripheral blood were collected from healthy control group, depression group and depression combined with cardiovascular disease group, and were analyzed by multi-omics. Subsequently, the patients were followed up in the outpatient clinic at 6 months, 1 year, 2 years and 5 years after discharge, and the clinical prognosis details of the patients were obtained and recorded.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
data of analysis of multi-omics | From enrollment to the end of five-year follow-up
  Samples of feces, urine and peripheral blood were collected from healthy control group, depression group and depression combined with cardiovascular disease group, and were analyzed by multi-omics. Subsequently, the patients were followed up in the outpatient clinic at 6 months, 1 year, 2 years and 5 years after discharge, and the clinical prognosis details of the patients were obtained and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided